CLINICAL TRIAL: NCT04402554
Title: Survey of Cannabis Use in Patients With Chronic Inflammatory Arthritis
Acronym: CannabisRIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 MATHIEU; 2020-A00473-36 (Other: 2020-A00473-36)
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Cannabis; Cannabis/therapeutic use; Cannabis/therapy; Medical Marijuana; Chronic Pain; Rheumatic Diseases; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Marijuana Abuse; Chronic Pain; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cannabis questionnaire — The effectiveness and use of cannabis in the management of chronic pain has been well known for many years, but has so far been illegal and therefore largely unacknowledged. We hypothesize that the use of cannabis in this population of patients with chronic joint or spinal pain is not anecdotal and responds to a need to further improve the overall management of patients. The objective of our anonymous questionnaire is to estimate the prevalence of cannabis use in patients with chronic inflammatory rheumatism.

SUMMARY:
Patients with inflammatory rheumatism very often have residual pain that is not easily relieved by conventional treatments. They can then use non-drug methods, such as physiotherapy, hypnosis or even cannabis.

The aim of this study is to assess the percentage of patients who use cannabis to better relieve their pain or anxiety in chronic inflammatory rheumatism.

DETAILED DESCRIPTION:
Thanks to a better understanding of the pathophysiological mechanisms of inflammatory rheumatism, rheumatology has known for several decades a growth in its therapeutic arsenal (csDMARDs, bDMARDs, tDMARDs). rheumatism control has thus been optimized.

however, patients very often keep pain, anxiety, residual fatigue, poorly controlled by our conventional therapies. patients then turn to non-drug therapies, among which the use of cannabis.

endocannabinoids have an analgesic and anti-inflammatory action recognized in pre-clinical trials. however, investigators currently lack the data to authorize its use in clinical rheumatology.

the aim of this study is to determine the prevalence of cannabis users in patients with rheumatoid arthritis, ankylosing spondyloarthritis or psoriatic arthritis in our unit. as a second intention, investigators will refine the consumption characteristics. Investigators will also look for possible risk factors for consumption (sensitivity to pain, catastrophism, standard of living, anxiety, depression, rheumatic activity and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis (ACR 2010 Criteria)
* Ankylosing Spondylitis (New york or ASAS criteria)
* Psoriatic Arthritis (CASPAR criteria)

Exclusion Criteria:

* Patient unable to complete questionnaires or unable to express informed consent
* Guardianship, trusteeship, deprivation of liberties, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Chronic Inflammatory Rheumatism, whether rheumatoid arthritis or spondyloarthritis, seen in consultation in the department of Rheumatology
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
prevalence of cannabis use in patients with chronic inflammatory rheumatic conditions | Day 0
  Patients will answer the following question: Are you currently using cannabis - Yes or No

SECONDARY OUTCOMES:
Percentage of patients with problematic cannabis use | Day 0
  Questionnaire CAST score. It includes 6 items with answer modes coded from 0 to 4. The total score obtained by summing these 6 items can therefore vary from 0 to 24. We define users without risk for a score of less than 3, users with low risk for a score greater than or equal to 3 and less than 7, and finally those with a risk of problematic use for a score greater than or equal to 7
Assessing the association between cannabis use and disease activity of spondylitis ankylosing | Day 0
  Spondylitis ankylosing activity was assessed by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questionnaire.
Assessing the association between cannabis use and disease activity of rheumatoid arthritis / psoriatic arthritis | Day 0
  Rheumatoid arthritis / psoriatic arthritis was assessed by Disease Activity Score including 28 joints (DAS 28). DAS 28 includes the 28 swollen joint count (28 SJC) + the 28 tender joint count (28 TJC) + patient global assessments of disease activity on a VAS, + ESR or CRP. [DAS (VS) = 0,56 x √TJC + 0,28 x √SJC + 0,7 x ln(VS) + 0,014 x VAS ; DAS (CRP) = 0,56 x √TJC + 0,28 x √SJC + 0,36 x ln(CRP + 1) + 0,014 x VAS + 0,96 ]. The scores according to EULAR criteria are: ≤2.6 for remission, >2.6 and ≤3.2 for low disease activity, >3.2 and ≤5.1 for moderate disease activity and >5.1 for high disease activity.
Assessing the association between cannabis use and functional disability | Day 0
  Functional disability was assessed by Health Assessment Questionnaire Disability Index (HAQ DI). HAQ-DI is an index that measures the impact of pathology on everyday activities such as dressing, eating, walking, etc.
  The following note is allocated to each question: 0 = without any difficulty ; 1 = with some difficulty ; 2 = with great difficulty ; 3 = unable to do so
Assessing the association between cannabis use and Anxiety/Depression | Day 0
  Anxiety and depression was assessed by Hospital Anxiety and Depression scale (HADs). 14 items scored from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing two scores to be obtained (maximum score of each score = 21). To detect anxious and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D): - 7 or less: absence of symptoms - 8 to 10: doubtful symptoms - 11 and more: certain symptoms.
Assessing the association between cannabis use and pain catastrophism | Day 0
  Catastrophism was assessed by Pain catastrophisme scale (PCS). PCS is a thirteen-item scale to identify and quantify the extent of catastrophism in a painful patient. Three subgroups group together the criteria related to rumination (items 8,9,10,11), exaggeration (items 6,7,13) and vulnerability (items 1,2,3,4,5,12) . Patients are asked to rate their personal experience using a five-point rating from 0 to 4. The final score can therefore vary from 0 to 52. A PCS score of 30 or more represents a relevant clinical level of catastrophism.
Assessing the association between cannabis use and social vulnerability | Day 0
  level of social vulnerability was assessed by Assessment of Precariousness and Health Inequalities in Health Examination Centers (EPICES) questionnaire.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Mathieu, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France